CLINICAL TRIAL: NCT05449587
Title: Study of the Long-Term Effectiveness of the Motiva Implants® Round and Round Ergonomix in Primary and Revision Breast Augmentation
Brief Title: Long-Term Effectiveness of the Motiva Implants® Round and Round Ergonomix
Acronym: MIRO
Status: Completed | Type: Observational
Sponsor: Motiva USA LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: CLINP- 001010
Record Dates: First submitted 2022-03-15; First posted 2022-07-08 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Breast Augmentation
Keywords: Revision Breast Augmentation; Primary Breast Augmentation; Breast Augmentation; Motiva Breast Implant; Silent rupture; Patient-Reported Outcomes
MeSH Terms: interventions — Magnetic Resonance Spectroscopy; prolyl-proline

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Primary /Revision Augmentation Cohort: Patients that underwent primary and/or revision augmentation from 3 years or more postoperatively.
  Interventions: Other: MRI and PRO

INTERVENTIONS:
Other: MRI and PRO — MRI as a standard of care for the analysis of silent rupture. BREAST-Q Postoperative Augmentation module scales to record patients for satisfaction: Satisfaction with breasts; Satisfaction with outcome; Psychosocial well-being; Physical well-being

SUMMARY:
Post-marketing surveillance study to demonstrate the silent rupture rate and satisfaction of patients who underwent a primary and revision breast augmentation surgery with Motiva Implants®, 3 to 10 years before enrollment.

DETAILED DESCRIPTION:
Single-arm, multicenter study with a minimum of 160 subjects who underwent Breast Implant surgery from 3-10 years postoperatively.

Following IRB / EC approval - and if applicable Competent Authority approval - Magnetic Resonance Imaging (MRI) and Patient-Reported Outcome (PRO) with the validated BREAST-Q will be collected at a single time point for all enrolled subjects.

MRI data will be used for the analysis of silent rupture, and BREAST-Q Postoperative Augmentation module scales to record patients for satisfaction.

Two styles of Motiva Implants® will be used for this study:

* Motiva Implants® Silicone Gel-Filled Breast Implants, SmoothSilk® Round (referred to as "Motiva Implants® Round ProgressiveGel® Plus", or "Round")
* Motiva Implants® Silicone Gel-Filled Breast Implants, SmoothSilk® Round Ergonomix® (referred to as "Motiva Implants® Ergonomix® Round ProgressiveGel® Ultima®", or "Round Ergonomix").

Henceforth, these devices will generally be referenced as "Motiva Implants®."

ELIGIBILITY:
Inclusion Criteria:

* Cisgender women.
* The subject has undergone primary or revision augmentation surgery with Motiva Implants® Round or Round Ergonomix®, which are still implanted before enrolling in the study.
* The subject underwent breast implant surgery at least three (3) years or more before enrolling in the study.
* The subject has undergone an MRI to evaluate implant rupture in the last 3 years before enrolling in the study or is willing to undergo an MRI evaluation.
* The subject is willing to follow all study requirements (signing informed consent, completing questionnaires, attending a baseline visit, and allowing access to previous MRI images or having new MRI images for the study).

Exclusion Criteria:

* The subject had undergone fat grafting, needle biopsy, or any procedures that might have caused an iatrogenic rupture.
* The Subject or Investigator are aware of a possible ruptured device that has not been removed.
* The subject is pregnant or nursing.
* The subject has any condition that impedes the use of Magnetic Resonance Imaging (MRI), including implanted metal devices, claustrophobia, or other conditions that would prohibit MRI scans.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Genetic women as inclusion criteria.
Study Population: Women who have undergone Primary/Revision Breast Augmentation with the Motiva Implants from 3 years or more postoperatively completed a breast MRI and the postoperative BREAST-Q Questionnaires.
Sampling Method: Non-Probability Sample
Enrollment: 111 (Actual)
Dates: Start 2022-11-22 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
To describe the rate of silent rupture in women who have undergone primary and revision breast augmentation with Motiva Implants® 3 to 10 years after surgery. | 1 year to complete after study start.
  Percentage of participants with silent implant rupture identified on MRI evaluation.
To describe Patient-Reported Outcomes in women who have undergone primary and revision breast augmentation with Motiva Implants® 3 to 10 years after surgery. | 1 year to complete after study start
  Mean scores of the BBREAST-QTM - AUGMENTATION MODULE (POSTOPERATIVE) VERSION 2.0, scales:
  * PSYCHOSOCIAL WELL-BEING. Values 1-5. A higher score means a better outcome.
  * SATISFACTION WITH BREASTS. Values 1-4. A higher score means a better outcome.
  * PHYSICAL WELL-BEING: CHEST. Values 1-3. A higher score means a worse outcome.
  * SATISFACTION WITH OUTCOME. Values 1-3. A higher score means a better outcome.

CONTACTS AND LOCATIONS:
Locations (2):
- Costa Rica (2):
  - Clinica de Cirugia Plastica Peralta Mantilla, Pavas, Provincia de San José
  - Centro Europeo de Cirugia, San José

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Calobrace MB, Schwartz MR, Zeidler KR, Pittman TA, Cohen R, Stevens WG. Long-Term Safety of Textured and Smooth Breast Implants. Aesthet Surg J. 2017 Dec 13;38(1):38-48. doi: 10.1093/asj/sjx157. PMID 29040370
- [Background] Zingaretti, Nicola & Fasano, Daniele & Preis, Franz & Moreschi, Carlo & Ricci, Silvia & Massarut, Samuele & De Francesco, Francesco & Parodi, Pier. (2020). Suspected breast implant rupture: our experience, recommendations on its management, and a proposal for a model of informed consent. European Journal of Plastic Surgery. 43. 10.1007/s00238-019-01610-1.
- [Background] Meadows KA. Patient-reported outcome measures: an overview. Br J Community Nurs. 2011 Mar;16(3):146-51. doi: 10.12968/bjcn.2011.16.3.146. PMID 21378658
- [Background] Wong T, Lo LW, Fung PY, Lai HY, She HL, Ng WK, Kwok KM, Lee CM. Magnetic resonance imaging of breast augmentation: a pictorial review. Insights Imaging. 2016 Jun;7(3):399-410. doi: 10.1007/s13244-016-0482-9. Epub 2016 Mar 9. PMID 26960549
- [Background] Ray JG, Vermeulen MJ, Bharatha A, Montanera WJ, Park AL. Association Between MRI Exposure During Pregnancy and Fetal and Childhood Outcomes. JAMA. 2016 Sep 6;316(9):952-61. doi: 10.1001/jama.2016.12126. PMID 27599330